CLINICAL TRIAL: NCT00850226
Title: Comparing Acceptance and Commitment Therapy Strategies to Cognitive Therapy Strategies in Reduction of Test Anxiety
Brief Title: Comparing Acceptance and Commitment Therapy (ACT) and Cognitive Therapy (CT) for Test Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Evan Forman, Ph.D., Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17111
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Anxiety
Keywords: test anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT (Experimental): Acceptance-and-Commitment Therapy Intervention: Subjects receiving the ACT strategies will be taught to defuse from their anxiety (or recognize that their thoughts are just thoughts). They will be taught to accept their anxiety and to learn to live with anxiety. Subjects will be told that while they cannot control the occurrence of their thoughts, they can control whether or not they choose to view them as separate from the self versus part of the self.
  Interventions: Behavioral: ACT
- CT (Experimental): Cognitive Therapy Intervention: Subjects receiving the CT strategies will be taught to restructure their negative thoughts to make them more positive, based on the concept that thoughts are linked to their problems with test anxiety because beliefs can cause strong powerful emotions and behaviors. Subjects will be taught not to blame their environments for emotional and behavioral responses, and they will be shown how to change their beliefs in order to affect their emotions and their behaviors.
  Interventions: Behavioral: CT

INTERVENTIONS:
Behavioral: CT — Cognitive Therapy Intervention: Subjects receiving the CT strategies will be taught to restructure their negative thoughts to make them more positive, based on the concept that thoughts are linked to their problems with test anxiety because beliefs can cause strong powerful emotions and behaviors. Subjects will be taught not to blame their environments for emotional and behavioral responses, and they will be shown how to change their beliefs in order to affect their emotions and their behaviors.
  Arms: CT
Behavioral: ACT — Acceptance-and-Commitment Therapy Intervention: Subjects receiving the ACT strategies will be taught to defuse from their anxiety (or recognize that their thoughts are just thoughts). They will be taught to accept their anxiety and to learn to live with anxiety. Subjects will be told that while they cannot control the occurrence of their thoughts, they can control whether or not they choose to view them as separate from the self versus part of the self.
  Arms: ACT

SUMMARY:
This study proposes to compare the effectiveness of an acceptance-based intervention and a cognitive control-based intervention for coping with test anxiety in nursing students during the HESI (Health Education Systems, Inc.) examination.

Subjects will be randomized to receive either the CT or the ACT condition. In both conditions, subjects will receive an education on test anxiety to inform them about what test anxiety is and why it occurs. Then, the different conditions will receive the respective treatment of either CT or ACT. The study is considered minimum risk because the nursing students will only be exposed to an amount of anxiety that is typical of their testing experience. Both conditions will meet three times, with each session lasting approximately one and a half hours. The purpose of the treatment is to provide subjects with tools to help them cope with their test anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Nursing student subjects may only participate if they are currently enrolled as an undergraduate student at Drexel University.
* They must be nursing majors enrolled in Nursing 492 and intending to take the cumulative HESI examination.
* Psychology students must be enrolled in the courses where recruitment will occur.
* Pre-professional students must be currently enrolled at Drexel University, and planning to take a Standardized test within 6 months.
* All subjects must be at least 18 years of age or older.

Exclusion Criteria:

* Persons may not participate if they are unable to see/read words off of a computer screen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
grades on final exams | 2-3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States